CLINICAL TRIAL: NCT02901418
Title: According to the Venous Blood HBsAg State of Neonatus at Birth, Discussing the Efficiency of Personalized Blocking Method of HBV Maternal-neonatal Transmission in High-risk Newborns
Brief Title: A Study of the Interruption on the Mother-to-child Transmission of Hepatitis B Virus （HBV MTCT）in Newborns at High Risk
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, Head of liver diseases center, Beijing Ditan Hospital
Other Study IDs: Z151122224015122
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Hepatitis B
Keywords: chronic hepatitis B; mother to child transmission; interruption; hepatitis B immunoglobulin; pregnancy; HBsAg; newborns
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — hepatitis B hyperimmune globulin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At the age of seven months, we extract venous blood of these children, separate the serums and collect the PBMC. Then, the serums are applied to test HBsAg, AntiHBs and HBVDNA which we adopt to analyse HLA classⅠand class Ⅱ gene polymorphism.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- control group: In this group,these children born in about two hours, we injected HBIG 200 iu and 10 micrograms of hepatitis b vaccine in their left and right thigh respectively, then injected 10 micrograms again in 1 and 6 months.
- experimental group: In this group,about 2 hours after birth, respectively injecting HBIG 200 IU and 10 micrograms of hepatitis b vaccine in the right and left thigh, and in 1 and 6 months again taking 10 micrograms of standard solution, in addition, offering the additional injection of 200 IU HBIG within 24 hours.
  Interventions: Biological: 200 IU HBIG

INTERVENTIONS:
Biological: 200 IU HBIG — additional 200 IU HBIG within 24 hours was used for the experimental group of newborns
  Other Names: hepatitis B immune globulin
  Groups: experimental group

SUMMARY:
Chronic hepatitis B (CHB) is a serious liver disease worldwide，HBV MTCT is the important reason to keep high prevalence of chronic HBV infection in China. Intrapartum infection is the main period of neonatal HBV infection. Injecting HBIG and hepatitis b vaccine immediately after birth is the most important method of blocking mother-to-child transmission of HBV. However, regular doses of HBIG combined with hepatitis b vaccine blocking measures still have a failure rate as high as 5% ~ 15%.There are numerous studies to explore pregnancy women with HBV positive, especially high viral load of those women during pregnancy being treated with nucleoside analogs to increase the blocking rate of HBV MTCT, but there is still a failure rate of 2.2% to 18%. In this study, we will explore the efficiency of personalized blocking method of HBV maternal-neonatal transmission in high-risk newborns,according to the venous blood HBsAg state of neonatus at birth.

DETAILED DESCRIPTION:
In this trial, the study population were consisted of patients suffering from chronic hepatitis B who had achieved HBeAg positive and HBV DNA > 106 copies/ml and their newborns who were born with HBsAg positive. Before injecting hepatitis b vaccine and HBIG for newborns, we tested their vein blood HBsAg levels, and the venous blood HBsAg positive newborns were randomly divided into the control group and the interventional group in which group we injected the additional 200 IU HBIG within 24 hours after birth, in addition to routine injection. We gathered the neonatal venous blood of 0, 7 and 30 days to test the level of anti HBs, HBsAg and HBV DNA., then detected the level of anti HBs, HBsAg and HBV DNA when these children were seven months.According to the venous blood HBsAg state of neonatus at birth, exploring the efficiency of personalized blocking method of HBV MTCT in high-risk newborns.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who were chronic hepatitis B and had achieved HBeAg positive and HBV DNA > 106 copies/ml
* At birth the neonatal venous blood HBsAg positive

Exclusion Criteria:

* Active consumption of alcohol and/or drugs
* Co-infection with human immunodeficiency virus, hepatitis C virus, or hepatitis D virus, HIV, etc.
* History of autoimmune hepatitis
* Psychiatric disease
* Evidence of neoplastic diseases of the liver
* without gestational hypertension, premature rupture of membranes, antepartum haemorrhage diseases or amniotic fluid piercing history during pregnancy.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: In this study,the study population were composed of pregnant women suffering from chronic hepatitis B who had achieved HBeAg positive and HBV DNA > 106 copies/ml and their newborns who were born with HBsAg positive
Sampling Method: Non-Probability Sample
Enrollment: 406 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
blocking rate of vertical transmission of hepatitis B | seven months
  At the birth of 7 months, the venous blood serum HBsAg positive was defined as the failure of the interruption of HBV mother-to-child transmission.

SECONDARY OUTCOMES:
anti HBs level at the age of one month and seven months | one month and seven months
  Observing the level of anti HBs, then discussing the efficiency of personalized blocking method of HBV maternal-neonatal transmission

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Ditan hospital,Capital Medical University, Beijing, Beijing Municipality, China